CLINICAL TRIAL: NCT06447324
Title: Assessment of Clinical, Radiographical Efficacy, Operator Ease and Satisfaction and Patient Comfort in Restoring Class II Cavities in Primary Molars With Fender Mate System Versus T-Band System: An in Vivo Study
Brief Title: Clinical and Radiographic Evaluation of Two Matrix Systems for Restoration of Class II Cavities in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Noha Elsayed Fathi Abdou, Lecturer at Pediatric Dentistry Department, Preventive Dentistry and Dental Public Health, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: matrix system for 1ry teeth
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Tooth Decay; Tooth Restoration
Keywords: Matrix Systems; Class II Cavities; Primary Molars
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: two groups
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fender Mate matrix group (Experimental): Twenty primary molars will be restored with composite restoration using the Fender Mate matrix
  Interventions: Device: Fender Mate matrix system
- Conventional T-band matrix group (Experimental): Twenty primary molars will be restored with composite restoration using T-band matrix
  Interventions: Device: T-band matrix

INTERVENTIONS:
Device: Fender Mate matrix system — Matrix Systems used for Restoration of Class II Cavities in Primary Molars
  Arms: Fender Mate matrix group
Device: T-band matrix — Matrix Systems used for Restoration of Class II Cavities in Primary Molars
  Arms: Conventional T-band matrix group

SUMMARY:
this study aims to evaluate and compare the clinical and radiographical efficacy, operator ease, satisfaction and patient comfort in restoring class II cavities in primary molars using Fender Mate system with T-band system.

DETAILED DESCRIPTION:
Restorations of posterior primary teeth can have a number of issues, including incorrect contact points and proximal overhangs. With the recognition of significance of restoring tooth's right contour and contact, and repair of all tooth surfaces, including proximal walls, different matrix systems were introduced,so this study aims to evaluate and compare the clinical and radiographical efficacy, operator ease, satisfaction and patient comfort in restoring class II cavities in primary molars using Fender Mate system with T-band system.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children free from any systemic diseases.
2. Patients showing Frankel's positive and definitely positive behavior.
3. Parent willing to participate in the study and signed on informed consent.
4. Each child has at least two carious primary molars (class II) bilaterally, indicated for composite restoration with criteria as follow: -

   * No history of spontaneous pain or provoked pain.
   * Fully erupted teeth.
   * Fully erupted adjacent tooth.
   * Caries involving two surfaces - proximal and occlusal
   * Absence of clinical signs or symptoms suggesting a non-vital tooth such as sinus tract, soft tissue swelling, mobility or tenderness to percussion.
   * No pathological external or internal root resorption.

Exclusion Criteria:

1. Patients showing Frankel's negative and definitely negative behavior.
2. Children having primary molars with:

   * Caries involving less than or more than two surfaces
   * Extensively damaged teeth
   * Missing adjacent tooth.
   * Mobility.
   * Spaced dentition.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of Proximal Contact Points | Baseline
  clinically assessment of the Proximal Contact Points using waxed dental floss in restoring class II cavities in primary molars using Fender Mate system in comparison with conventional T-band matrix.
Radiographically Assessment of proximal overhangs | Baseline
  Radiographically Assessment of the proximal overhangs using bite wing radiograph in restoring class II cavities in primary molars using Fender Mate system in comparison with conventional T-band matrix.
Assessment of operator ease and satisfaction | Baseline
  -Assessment of operator ease and satisfaction using questionnaire in restoring class II cavities in primary molars using Fender Mate system in comparison with conventional T-band matrix, which includes:
  1. time needed to install the matrix system (more time means worse outcome)
  2. Ease of application and removal of matrix system which may be Easy, Manageable or Difficult (Difficult means worse outcome)
  3. Trauma to gingival tissue while applying and removing matrix system which may be Present or Absent (Present means worse outcome)
  4. Dislodgment/displacement of restoration while removing matrix system which may be Yes or NO (Yes means worse outcome)
Assessment of patient comfort | Baseline
  * Assessment of patient comfort using Wong Baker pain rating scale in restoring class II cavities in primary molars using Fender Mate system in comparison with conventional T-band matrix.
  * Wong Baker pain rating scale with scores from 0-10 (higher scores mean a worse outcome).

REFERENCES:
- [Result] Dindukurthi MK, Setty JV, Srinivasan I, Melwani AM, Manasa Hegde K, Radhakrishna S. Restoration of Proximal Contacts in Decayed Primary Molars Using Three Different Matrix Systems in Children Aged 5-9 Years: An In Vivo Study. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):70-74. doi: 10.5005/jp-journals-10005-1929. PMID 34326587
- [Result] Bhatia HP, Sood S, Sharma N, Singh A, Rajagopal V. Comparative Evaluation of Clinical Efficiency and Patient Acceptability toward the Use of Circumferential Matrix and Sectional Matrix for Restoration of Class II Cavities in Primary Molars: An In Vivo Study. Int J Clin Pediatr Dent. 2021 Nov-Dec;14(6):748-751. doi: 10.5005/jp-journals-10005-2060. PMID 35110865
- [Result] Gomes IA, Filho EM, Mariz DC, Borges AH, Tonetto MR, Firoozmand LM, Kuga CM, De Jesus RR, Bandeca MC. In vivo Evaluation of Proximal Resin Composite Restorations performed using Three Different Matrix Systems. J Contemp Dent Pract. 2015 Aug 1;16(8):643-7. doi: 10.5005/jp-journals-10024-1735. PMID 26423500